CLINICAL TRIAL: NCT05645107
Title: A Randomized, Multi-Center, Parallel, Double-Blinded, Placebo-Controlled Clinical Trial to Evaluate Efficacy, Safety, and Pharmacokinetics of XEMBIFY® Plus Standard Medical Treatment Compared to Placebo Plus Standard Medical Treatment to Prevent Infections in Patients With Hypogammaglobulinemia and Recurrent or Severe Infections Associated With B-cell Chronic Lymphocytic Leukemia, Multiple Myeloma, and Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate Efficacy, Safety, and PK of XEMBIFY®+Standard Medical Treatment (SMT) Compared to Placebo+SMT to Prevent Infections in Participants With HGG and Recurrent or Severe Infections Associated With B-cell Chronic Lymphocytic Leukemia, Multiple Myeloma, and Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GC2202; XEMBIFY® - CLL, MM, and NHL (Other: Grifols Therapeutics LLC); 2022-502193-16-00 (Other: EU CT)
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hypogammaglobulinemia; Bacterial Infections; B-cell Chronic Lymphocytic Leukemia; Multiple Myleoma; Non-Hodgkin Lymphoma
Keywords: XEMBIFY; CLL; SMT; Hypogammaglobulinemia (HGG); MM; NHL
MeSH Terms: conditions — Agammaglobulinemia; Bacterial Infections; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — gamma-Globulins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XEMBIFY + Standard Medical Treatment (SMT) (Experimental): Participants will receive a loading dose of 150 milligrams per kilograms per day (mg/kg/day) (Week 1, Days 1 to 5) subcutaneously (SC) for 5 consecutive daily doses followed by biweekly infusions of 300 mg/kg/2-week starting Week 3 (Day 15) through Week 51 (end of Treatment Phase).
  The SMT will include the active treatments and the other supportive treatments that the participants will need during their participation.
  Interventions: Drug: Xembify
- Placebo + SMT (Placebo Comparator): Participants will receive sterile 0.9 percent Sodium Chloride Injection (commercially available in the corresponding country) starting at Week 1 (Days 1 to 5) SC for 5 consecutive daily doses followed by biweekly infusions starting at Week 3 (Day 15) through Week 51.
  The SMT will include the active treatments and the other supportive treatments that the participants will need during their participation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xembify — SC infusion pump
  Other Names: Immune Globulin Subcutaneous (Human), 20% (IGSC 20%)
  Arms: XEMBIFY + Standard Medical Treatment (SMT)
Drug: Placebo — SC infusion pump
  Other Names: 0.9% Normal Saline
  Arms: Placebo + SMT

SUMMARY:
The primary purpose of the study is to evaluate whether biweekly administered XEMBIFY® plus Standard Medical Treatment (SMT) over a one-year period will reduce the rate of major bacterial infections per participant per year in B-cell CLL, MM, and NHL participants with hypogammaglobulinemia (HGG) in comparison to the Placebo plus SMT group.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age at screening visit
* Participants with documented and confirmed diagnosis of any of the below diseases:

  * B-cell CLL according to International Workshop on CLL (iwCLL) criteria and RAI staging of intermediate (1 and 2) or high (3 and 4)
  * MM according to the International Myeloma Working Group criteria (IMWG), R-ISS stage II or, III; or
  * Histologically confirmed diagnosis of B-Cell NHL, Stage III or above (IV, Progressive/refractory, or recurrent/relapsed stage) according to the Lugano Classification.
* Participants with HGG with IgG levels less than 5 g/L.
* Participants with documented history of at least one severe bacterial infection (bacterial or viral) or recurrent bacterial/viral infections (that is., ≥ 3 infections) within 12 months before the screening visit. Severe bacterial/viral infections ≥ Grade 3 (as defined by Common Terminology Criteria for Adverse Events [CTCAE] Grades).

Exclusion Criteria:

* Participants with documented history of hematopoietic stem cell transplant.
* Participants currently receiving immunoglobulin replacement therapy (IgRT) or have received IgG replacement treatment (i.e., prior immune globulin replacement therapy) within 6 months before the screening visit.
* Participants with active infections at time of screening visit. Specific supportive anti-infective prophylactic defined in the CLL National Comprehensive Cancer Network (NCCN) or iwCLL guidelines and/or local/international guidelines for the CLL, and defined in local/international guidelines for MM and NHL are allowed, or recommended in the updated labelling of specific active target disease medicines used during the participation in the trial is also allowed.
* Participants with active second malignancies.
* Participants with known primary immunodeficiency (PI).
* Participants with a life expectancy less than 1.5 years.
* Participants with clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may interfere with successful completion of the trial or place the subject at undue medical risk.
* Participants have had a known serious adverse reaction (AR) to immunoglobulin or any anaphylactic reaction to blood or any blood-derived product.
* Participants have a history of blistering skin disease, bleeding disorder, diffuse rash, recurrent skin infections, or other disorders where SC therapy would be contraindicated during the study based upon the Investigator's discretion.
* Participants have known Selective Immunoglobulin A (IgA) Deficiency (with or without antibodies to IgA) (Note: exclusion is for the specific diagnostic entity. It does not exclude other forms of humoral primary immunodeficiency which have decreased IgA in addition to decreased IgG requiring IgG replacement).
* Participants with severe known kidney disease [as defined by estimated glomerular filtration rate [eGFR] less than (<) 30 milliliter (mL)/min/1.73 square meter (m2)] as determined by the Principal Investigator.
* Participants that have liver enzyme levels (alanine aminotransferase [ALT], aspartate aminotransferase [AST], gammaglutamyl transferase [GGT], or lactate dehydrogenase [LDH]) greater than 3 times the upper limit of normal (ULN) at the Screening Visit as defined by the testing laboratory.
* Participants have a history (either 1 episode within the year prior to the Screening Visit or 2 previous episodes over a lifetime) of or current diagnosis of thromboembolism (example, myocardial infarction, cerebrovascular accident, or transient ischemic attack) or deep venous thrombosis.
* Participants currently have a known hyperviscosity syndrome or hypercoagulable states.
* Participants have a known previous infection or clinical signs and symptoms consistent with current hepatitis B virus or hepatitis C virus infection.
* Participants with non-controlled arterial hypertension (systolic blood pressure [SBP] greater than 140 millimeters of mercury (mmHg) and/or diastolic blood pressure [DBP] greater than 90 mmHg), and/or a heart rate (HR) greater than100 bpm.
* Participants with known substance or prescription drug abuse within 12 months before the Screening Visit.
* Participants have participated in another clinical trial within 30 days prior to screening (observational studies without investigative treatments [non-interventional] are permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Annual Rate of Major Bacterial Infections per Year | Up to Week 51

SECONDARY OUTCOMES:
Time to First Onset of Major Bacterial Infection | Up to Week 51
Percentage of Participants who Experience Major Bacterial Infections | Up to Week 51
Rate of all Bacterial Infections Determined by the Investigator | Up to Week 51
Percentage of Participants who Experience Bacterial Infections | Up to Week 51
Time to First Onset of Non-Major Bacterial Infections | Up to Week 51
Number of Days on Which Participants Were on Antibiotics | Up to Week 51
Number of Hospitalizations due to any Infections | Up to Week 51
Duration of Hospitalizations due to any Infections | Up to Week 51
Number of Hospitalizations due to Major Bacterial Infections | Up to Week 51
Duration of Hospitalizations due to Major Bacterial Infections | Up to Week 51
Rate of all Infections as Determined by the Investigator | Up to Week 51
Number of Participants with Validated Infections | Up to Week 51
Time to First Onset of any Infection | Up to Week 51

CONTACTS AND LOCATIONS:
Locations (59):
- United States (6):
  - GC2202 Study Site 103, St. Petersburg, Florida
  - GC2202 Study Site 111, Bethesda, Maryland
  - GC2202 Study Site 109, Greenville, North Carolina
  - GC2202 Decentralized Study Site 114, Morrisville, North Carolina
  - GC2202 Study Site 105, Canton, Ohio
  - GC2202 Study Site 110, Rockville, South Carolina
- Bosnia and Herzegovina (3):
  - GC2202 Study Site 702, Banja Luka
  - GC2202 Study Site 703, Mostar
  - GC2202 Study Site 701, Sarajevo
- Bulgaria (14):
  - GC2202 Study Site 202, Burgas
  - GC2202 Study Site 203, Plovdiv
  - GC2202 Study Site 210, Plovdiv
  - GC2202 Study Site 205, Rousse
  - GC2202 Study Site 209, Sofia
  - GC2202 Study Site 201, Sofia
  - GC2202 Study Site 206, Sofia
  - GC2202 Study Site 207, Sofia
  - GC2202 Study Site 211, Sofia
  - GC2202 Study Site 212, Sofia
  - GC2202 Study Site 213, Sofia
  - GC2202 Study Site 204, Sofia
  - GC2202 Study Site 208, Sofia
  - GC2202 Study Site 214, Stara Zagora
- Croatia (2):
  - GC2202 Study Site 801, Rijeka
  - GC2202 Study Site 802, Zagreb
- Hungary (8):
  - GC2202 Study Site 305, Székesfehérvár, Fejér
  - GC2202 Study Site 301, Budapest
  - GC2202 Study Site 308, Budapest
  - GC2202 Study Site 306, Debrecen
  - GC2202 Study Site 304, Eger
  - GC2202 Study Site 302, Győr
  - GC2202 Study Site 307, Szeged
  - GC2202 Study Site 303, Szekszárd
- Poland (9):
  - GC2202 Study Site 402, Torun, Kuyavian-Pomeranian Voivodeship
  - GC2202 Study Site 401, Krakow, Lesser Poland Voivodeship
  - GC2202 Study Site 403, Legnica, Lower Silesian Voivodeship
  - GC2202 Study Site 406, Wałbrzych, Lower Silesian Voivodeship
  - GC2202 Study Site 405, Słupsk, Pomeranian Voivodeship
  - GC2202 Study Site 408, Bydgoszcz
  - GC2202 Study Site 410, Krakow
  - GC2202 Study Site 409, Olsztyn
  - GC2202 Study Site 407, Torun
- Romania (10):
  - GC2202 Study Site 503, Brasov, RO
  - GC2202 Study Site 504, Bucharest, RO
  - GC2202 Study Site 506, Cluj-Napoca, RO
  - GC2202 Study Site 502, Timișoara, RO
  - GC2202 Study Site 509, Bucharest
  - GC2202 Study Site 511, Bucharest
  - GC2202 Study Site 508, Bucharest
  - GC2202 Study Site 501, Bucharest
  - GC2202 Study Site 507, Constanța
  - GC2202 Study Site 510, Iași
- Serbia (7):
  - GC2202 Study Site 602, Belgrade
  - GC2202 Study Site 604, Belgrade
  - GC2202 Study Site 605, Belgrade
  - GC2202 Study Site 607, Belgrade
  - GC2202 Study Site 603, Kamenitz
  - GC2202 Study Site 601, Kragujevac
  - GC2202 Study Site 606, Niš

IPD SHARING:
Plan to Share IPD: No